CLINICAL TRIAL: NCT01134523
Title: Phase 3 Study of Regimens Comparison for Breast Cancers of Positive Lymph Nodes
Brief Title: Regimens Comparison for Breast Cancers of Positive Lymph Nodes
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Binghe Xu, Chief, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CH-BC-006
Record Dates: First submitted 2010-06-01; First posted 2010-06-02 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Breast Cancer
Keywords: positive lymph node
MeSH Terms: conditions — Breast Neoplasms | interventions — Epirubicin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A: EC-T regimen (Active Comparator)
  Interventions: Drug: Epirubicin, CTX, Paclitaxel
- Group B: ET regimen (Experimental)
  Interventions: Drug: Epirubicin, Paclitaxel

INTERVENTIONS:
Drug: Epirubicin, CTX, Paclitaxel — Epirubicin 90mg/m2 and CTX 600mg/m2 on day1 of each 21-day cycle, 4 cycles; followed by Paclitaxel 175mg/m2 on day1 of each 21-day cycle, 4 cycles.
  Arms: Group A: EC-T regimen
Drug: Epirubicin, Paclitaxel — Epirubicin 75mg/m2 on day1 and Paclitaxel 175mg/m2 on day2 of each 21-day cycle, 6 cycles.
  Arms: Group B: ET regimen

SUMMARY:
To compare the efficacy and safety of EC-T and ET regimen as adjuvant treatment of breast cancer patients with positive lymph nodes

DETAILED DESCRIPTION:
EC-T regimen: epirubicin 90mg/m2 day1, CTX 600mg/m2, day 1, 21 days per cycle *4cycle. followed by paclitaxel 175mg/m2,d1,21days per cycle, 4 cycle.

ET regimen: epirubicin 75mg/m2 day1,paclitaxel 175mg/m2,d2,21days per cycle, 6 cycle

ELIGIBILITY:
Inclusion Criteria:

* patients with breast cancer after breast cancer surgery with positive lymph nodes age 18-70 years old

Exclusion Criteria:

* with other malignance disease

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2010-05; Primary Completion 2018-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
PFS | 5 years after all the recuiment

SECONDARY OUTCOMES:
OS | 5 years after all the adjuvent treatments
Safety | 5 years after all the recruiment
  Assessing for Hematology and Non-hematology toxicities, including all SAEs.

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, M.D., Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute & Hospital. Chinese Academy of Medical Sciences, Beijing, China

REFERENCES:
- [Background] Moebus V, Jackisch C, Lueck HJ, du Bois A, Thomssen C, Kurbacher C, Kuhn W, Nitz U, Schneeweiss A, Huober J, Harbeck N, von Minckwitz G, Runnebaum IB, Hinke A, Kreienberg R, Konecny GE, Untch M. Intense dose-dense sequential chemotherapy with epirubicin, paclitaxel, and cyclophosphamide compared with conventionally scheduled chemotherapy in high-risk primary breast cancer: mature results of an AGO phase III study. J Clin Oncol. 2010 Jun 10;28(17):2874-80. doi: 10.1200/JCO.2009.24.7643. Epub 2010 May 10. PMID 20458045
- [Derived] Yuan P, Kang Y, Ma F, Fan Y, Wang J, Wang X, Yue J, Luo Y, Zhang P, Li Q, Xu B. Effect of Epirubicin Plus Paclitaxel vs Epirubicin and Cyclophosphamide Followed by Paclitaxel on Disease-Free Survival Among Patients With Operable ERBB2-Negative and Lymph Node-Positive Breast Cancer: A Randomized Clinical Trial. JAMA Netw Open. 2023 Feb 1;6(2):e230122. doi: 10.1001/jamanetworkopen.2023.0122. PMID 36826820
- See also: http://www.ncbi.nlm.nih.gov/pubmed/20458045 — http://www.ncbi.nlm.nih.gov/pubmed/20458045